CLINICAL TRIAL: NCT03213600
Title: Neurostimulation-enhanced Behavioral Remediation of Social Cognition in Schizophrenia
Acronym: NSOCOG
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: One of the investigators went abroad
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2017-A01042-51
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Behaviors and Mental Disorders
MeSH Terms: conditions — Behavior; Mental Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: The investigators will enroll 150 subjects comprising three population groups SZ, At Risk and HS.) Immediately after inclusion, participants will be randomized into 2 equal groups via random generation of two binary integer's reflecting tDCS-treatment condition or the tDCS control (sham) resulting in random allocation into one of 2 study arms. This randomization will be stratified per population group to insure that both conditions are equally reflected across all three groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transcranial Direct Current Stimulation ( tDCS ) (Active Comparator): Intensity : 1,5mA Duration : 20 minutes stimulation over frontal (F3/F4) electrodes
  Interventions: Device: transcranial Direct Current Stimulation tDCS
- transcranial Direct Current Stimulation ( tDCS) (Sham Comparator): Intensity : 1,5mA Duration : 20 minutes stimulation over parietal(CP3 CP4) electrodes
  Interventions: Device: transcranial Direct Current Stimulation tDCS

INTERVENTIONS:
Device: transcranial Direct Current Stimulation tDCS — 75 participants will receive 20 minutes of active tDCS (1,5mA, 20 minutes stimulation over frontal (F3/F4) electrodes ); A group of 75 participants will receive 1,5mA 20 minutes of stimulation over parietal (CP3 CP4) electrodes. During this stimulation session and we will also measure your ability to perceive visual and auditory objects presented by a computer, while recording your brain activity using electroencephalography or EEG (a technique using electrodes that measures the electrical activity of your brain)

SUMMARY:
Social cognition concerns the understanding of how people think about others and how that, in turn, influences our behavior, feelings, and social interactions. schizophrenia social-cognitive impairment is profound (effect size D>1.2), medication resistant and critically limits functional well-being . Social cognition involves complex patterns of coordinated activity within numerous cortical and subcortical networks, making it a difficult target for clinical neuroscience investigation. Yet, prior research demonstrates that sensory-perceptual dysfunction in schizophrenia can upwardly generalize into higher-order social-cognitive impairment making perception a tractable and fruitful approach for studying social cognition in schizophrenia. Here, the investigators explore how distortions in perception of temporal coincidence can contribute to the aberrant inferences of physical causation and social agency.

DETAILED DESCRIPTION:
Social cognitive deficits in these patients are robust and hinder their ability to maintain gainful employment as well as forge and sustain meaningful social relationships. Current antipsychotic medications are largely ineffective in treating these symptoms. The proposed protocol aims at utilizing Noninvasive Brain Stimulation (NIBS) and cognitive behavioral training to enhance core perceptual impairment in marking time that may contribute to both social and nonsocial cognitive dysfunction in schizophrenia.

Cognitive behavioral training along the line investigators propose has no reported adverse effects.The transdirect current stimulation (tDCS) is a very safe method with encouraging results in previous works in which no severe adverse events where found. There are a few minor side effects including skin irritation, a phosphene at the start of stimulation, nausea, headache, dizziness, and itching under the electrode. A recent study of over 500 subjects using the currently accepted protocol reported only a slight skin irritation and a phosphene as side effects. Patients can benefit from a significant improvement of invalidant symptoms but also of their quality of life. To ensure safety, patients will be accompanied throughout the protocol by professionals trained in the management of their disease. Besides the protocol procedure, patients will be supported, in all centers, according to the international recommendations in terms of safety and practice. Patients receiving placebo procedure after randomization will pursue pharmacological treatment and usual health care.

ELIGIBILITY:
Inclusion Criteria:

* be between 18 and 45-years-old
* have normal hearing assessed by the Five-minute hearing test
* have French as a first language
* be able to provide written informed consent
* be right handed as measured by the Edinburgh handedness scale
* covered by, or having the right to Social Security
* informed consent signed
* patients with diagnosis of schizoprenia or schizoaffective disorder-depressive type as determined by the SCID Diagnostic Interview for DSM-V and administered by a clinician
* clinically stable and on a stable medication regiment for the past 3 months

Exclusion Criteria:

* significant medical or neurological illness or history of fetal alcohol exposure that may increase risks of the study, significantly affect brain function, or impede participation
* substance dependence (except nicotine) or abuse not in remission within the past six months or recent use presenting the possibility of acute intoxication or withdrawal
* a history of any Axis I psychiatric disorder except those required in the inclusion criteria, any history of pervasive developmental disorder or mental retardation
* for Visit 3: If participating in tCDS Contraindications for tDCS (pacemaker or brain stimulator) and/or MRI (neurologic stimulator, pacemaker, cardiac defibrillator, cardiac prosthesis, vascular prosthesis, intracranial clips or clamps, cerebrospinal fluid derivation, metallic splinters in the eyes)
* patients under curatorship/guardianship and whose clinical condition requires inpatient procedure under constraint
* healthy controls must not be currently using psychoactive médications or have a first-degree relative with a psychotic disorder

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Causation Task - testing time based causal judgments | 3 months
  Primary metric: threshold defined as the smallest time difference (in 16.7ms increments) at which subject judge ball movement "B" to be caused by the impact of ball "A" 75% of the time.
Triangle Task - measuring the extent to which temporal coincidence is used to infer causality in a social situation | 3 months
  Primary metric: threshold of tolerated relational time delay (levels in 16.7ms increments) between interacting visual figures (i.e triangles), under which participants reliably (at 75%) perceive social agency or social interactions.

SECONDARY OUTCOMES:
EEG Task 1, Time visual oddball task - for measuring electrophysiological markers of active temporal (time) deviance detection | 3 months
  Primary metric: Mismatch negativity in the event related potentials of electrodes over the visual cortex with typical latency of 150-250ms after the onset of the deviant stimuli
EEG Task 2, Covert visual simultaneity task - an exploratory task designed to model the visual Simultaneity behavioral task | 3 months
  Primary metric: Dependent measure: decibel change in Alpha and Beta power across bellow- threshold and above- threshold conditions
Resting state oscillatory structure | 3 months
  Primary metric: Dependent measure: decibel change in Alpha and Beta power during rest

CONTACTS AND LOCATIONS:
Overall Officials: POULET EMMANUEL, MD - PhD, Principal Investigator — CH LE VINATIER
Locations (1):
- Hopital Le Vinatier, Bron, France